CLINICAL TRIAL: NCT06501742
Title: Major Hepatectomy and Vascular Clamping: Pre- and Intra-operative Predictive Factors of Vascular Clamping, Intra- and Post-operative Tolerance
Brief Title: Major Hepatectomy and Vascular Clamping
Acronym: HMCV
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9138
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Liver Diseases
Keywords: Liver Diseases; Hepatectomy; Liver Cancer
MeSH Terms: conditions — Liver Diseases; Liver Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A major hepatectomy consists of the resection of 3 or more liver segments. Its indications are mainly secondary malignant lesions, then primary malignant lesions, benign lesions and septic resections. Around a hundred major hepatectomies are carried out every year in Strasbourg. This surgery is burdened by 4.5% mortality at day 90 and 20 to 50% morbidity. The main intraoperative risks are hemorrhage and hemodynamic instability. Surgical vascular clamping helps reduce the risk of bleeding but is responsible for sometimes major hemodynamic variations, ischemia-reperfusion syndromes and can lead to acute post-operative liver failure. Recent literature attests to the safety of liver resection without vascular clamping, which is why it is less and less practiced.

Different elements are identified as independent risk factors for morbidity and mortality: the presence of cirrhosis, portal embolization, history of renal or cardiac failure, duration of vascular clamping, resected liver volume, transfusion of products labile blood and associated surgical procedures.

Given the significant risk of intra- and post-operative complications, it seems relevant to analyze pre- and intra-operative data in order to highlight risk factors for vascular clamping. This would allow better anticipation of complications, patient information, adaptation of intraoperative monitoring and postoperative surveillance and perhaps a reduction in complications. This study also makes it possible to take stock of the epidemiology around hepatectomies performed at the STRASBOURG University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Major subject (≥ 18 years old)
* Subject operated on for a major hepatectomy at Strasbourg University Hospital during the period from January 1, 2023 to December 31/2023
* Subject who has not expressed opposition to the reuse of their data for scientific research purposes.

Exclusion Criteria:

* Subject having expressed opposition to participating in the study
* History of liver resection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subject (≥ 18 years old) operated on for a major hepatectomy at Strasbourg University Hospital during the period from January 1, 2023 to December 31/2023
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Analyze pre- and intra-operative data from a major hepatectomy in order to identify possible predictive factors for intra-operative vascular clamping. | Up to 1 year
  Quantitative variables are described using the usual position and dispersion statistics, namely mean, median, minimum, maximum, standard deviation and quantile. The qualitative variables are described with the numbers (in number) and proportions (in %)of each modality.
  The Chi2 test will be used to study the crossover between

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Anesthésie - Réanimation Chirurgicale - CHU de Strasbourg - France, Strasbourg, France